CLINICAL TRIAL: NCT05728372
Title: Pilot Trial Using 64Cu-DOTA Pembrolizumab (64CDP) in Patients Receiving Stereotactic Body Radiation Therapy for Oligo-Progressive Solid Tumors
Brief Title: 64Cu-DOTA Pembrolizumab for Imaging Metastatic Solid Tumors in Patients Receiving Stereotactic Body Radiation
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: withdrawn per PI
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22305; NCI-2022-10254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22305 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-02-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (64CDP PET) (Experimental): Patients receive standard of care pembrolizumab IV at baseline. Patients then receive 64CDP IV days 1 and 29 on study. Patients undergo PET scan on days 2 and 30 on study. Patients also undergo standard of care SBRT days 8-18.
  Interventions: Drug: Copper Cu 64-DOTA-pembrolizumab; Procedure: Positron Emission Tomography; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Copper Cu 64-DOTA-pembrolizumab — Given IV
  Other Names: 64Cu-DOTA-pembrolizumab; 64Cu-labeled Pembrolizumab; 64Cu-pembrolizumab; Copper Cu 64 Pembrolizumab
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This clinical trial tests how well using 64Cu-DOTA pembrolizumab (64CDP) with positron emission tomography (PET) scans works to find tumor cells in patients with cancers that have spread from where it first started to other places in the body (metastatic). 64CDP is a compound with pembrolizumab that is joined with a radioactive substance used for diagnostic purpose. Pembrolizumab is in a class of medications called monoclonal antibodies. It works by helping your immune system to slow or stop the growth of cancer cells. Targeted drugs such as pembrolizumab may the improve uptake of the radioactive substance in tumor cells. 64CDP may improve ability to evaluate response to treatment in patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe toxicities of 64Cu-DOTA-pembrolizumab (64CDP) positron emission tomography, by evaluation of toxicities including: type, frequency, severity, attribution, time course, and duration.

II. To identify changes in 64Cu-DOTA-pembrolizumab (64CDP) uptake in radiated metastatic lesions pre- and post-SBRT.

OUTLINE:

Patients receive standard of care pembrolizumab intravenously (IV) at baseline. Patients then receive 64CDP IV days 1 and 29 on study. Patients undergo PET scan on days 2 and 30 on study. Patients also undergo standard of care SBRT days 8-18.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: >= 18 years
* Karnofsky performance status (KPS) >=70
* Patients with metastatic disease from a solid-tumor malignancy currently being treated with single-agent pembroilizumab, who have been referred for stereotactic body radiation therapy (SBRT) for consolidative local therapy or for oligo resistant/progressive disease
* Sites that amenable to SBRT are located in lymph nodes, bone/spine, or lung
* Brain metastases or cases with intra-cranial progression are allowed, but an additional extra-cranial site planned for SBRT is required
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 50/mm^3; platelet transfusions to help patients meet eligibility criteria are not allowed within 7 days before study enrollment
* Total bilirubin =< 1.5 x the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Calculated creatinine clearance >= 30mL/min
* Contraception:

  * Woman of childbearing potential must be practicing a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods; condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization; true abstinence (when this is in line with the preferred and usual lifestyle of the subject) during and after the study (6 months after the last dose of 64Cu-anti-PD1 [pembrolizumab]-NHS-DOTA for women);
  * A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control, e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 6 months after receiving the last dose of study drug

Exclusion Criteria:

* Patient planned to stop Pembrolizumab at time of referral for SBRT
* Patient unable to tolerate positron emission tomography (PET) scan even with anxiolytic medications
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Vaccination with live attenuated vaccines within 4 weeks of study agent administration except forthcoming COVID-19 vaccines
* Subject is currently using or has used immunosuppressive medication within 14 days prior to the study agent administration with the exception of:

  * Intranasal, topical, inhaled, or local steroid injections (e.g., intra-articular injection);
  * Chronic systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., infusion-related reactions, CT scan premedication)
* Female patients who are lactating or have a positive pregnancy test during the screening period
* Infection requiring systemic antibiotic therapy within 14 days prior to start of study treatment
* Subject has plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or primary amyloidosis
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-25 (Estimated); Primary Completion 2026-11-08 (Estimated); Study Completion 2026-11-08 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | After administration of study treatment up to 1 month
  Defined as any infusion-related reactions, hematologic or non-hematologic toxicities that occur during the first 3 days post administration of study drug that are possibly related to protocol therapy. DLT adverse events will be monitored continuously. Toxicities will be summarized in terms of type, severity, time of onset, duration, and association with study treatment.
Changes in 64CDP uptake | From baseline through study completion, an average of 6 weeks
  T-test to determine significance. T-tests (paired) will be used to test changes in 64-CDP uptake in radiated metastatic lesions pre- and post-SBRT.
Change in standard-uptake-value (SUV-max) | From baseline through study completion, an average of 6 weeks
  T-test to determine significance.
Incidence of adverse events | After administration of study treatment up to 1 month
  Defined as any infusion-related reactions, hematologic or non-hematologic toxicities that occur during the first 3 days post administration of study drug that are possibly related to protocol therapy. Dose limiting toxicity (DLT) adverse events will be monitored continuously. Toxicities will be summarized in terms of type, severity, time of onset, duration, and association with study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sagus Sampath, Principal Investigator — City of Hope Medical Center